CLINICAL TRIAL: NCT00632307
Title: Detection of Clusters of Volatile Organic Compounds (VOC)in Patients With Different Lung Disorders by Ion Mobility Spectrometry. Different Clusters of VOC in the Diagnosis of Different Lung Disorders Using Ion Mobility Spectrometry
Brief Title: Breath Analysis by Ion Mobility Spectrometry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lung Clinic Hemer (Other)
Responsible Party: Principal Investigator, Michael Westhoff MD, Dr. Michael Westhoff, Lung Clinic Hemer
Other Study IDs: lkhemer1-2008
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Lung Diseases
Keywords: lung tumor; pleural tumor; interstitial lung disease; airway infection; COPD; sleep apnea; ion mobility spectrometry; breath analysis
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms; Pleural Neoplasms; Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — breath, pleural fluid (only in patients with therapeutic pleurocentesis)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- 1: COPD
- 2: lung cancer
- 3: airway infection
- 4: interstitial lung disease
- 5: sleep apnea
- 6: pulmonary disorders with pleural infusions
- 7: sarcoidosis
- 8: healthy persons

SUMMARY:
Recognition of disease specific clusters of volatile organic compounds in patients with different lung diseases, using breath analysis with ion mobility spectrometry. Lung diseases of interest are:

* COPD
* tumors
* airway infection
* interstitial lung disease
* sleep apnea Hypothesis: Breath analysis with ion mobility spectrometry can differentiate pulmonary disorders.

DETAILED DESCRIPTION:
Recruitment of patients with different lung diseases goes on. First sub-group analysis of patients with COPD,lung cancer and sarcoidosis is done in order to create a training set of VOC-clusters for further validation in a bigger population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patient
* Ages 18-90 years old

Exclusion criteria:

- Patient who are not able to perform an exhalation manoever.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients of the lung clinic hemer with pulmonary diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-07; Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of diseases specific VOCs | years

SECONDARY OUTCOMES:
Change of disease specific VOCs under therapy | years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Westhoff, MD, Principal Investigator — Lung Clinic Hemer, 58675 Hemer, Germany
Locations (1):
- Lung Clinic Hemer, Hemer, Germany

REFERENCES:
- [Background] Westhoff, M; Litterst, P; Bödeker, B; Baumbach, J: Beath analysis by IMS for differentiation of COPD und Interstitial Lung Disease Pneumologie; 2011, 65: P278
- [Background] Westhoff, M; Litterst, P; Madulla S, Bödeker, B; Baumbach, J Differentiation of COPD patients including patients with lung cancer from healthy persons by IMS. Implementation of statistic and bioinformatic methods. Pneumologie 2012; 66: V394
- [Background] Westhoff M, Litterst P, Maddula S, Baumbach JI Differentiation of chronic obstructive pulmonary disease (COPD) including lung cancer from healthy control group by breath analysis using ion mobility spectrometry Eur Respir J 2011; 38: Suppl 55, P1699
- [Background] Westhoff M, Litterst P, Sommer H, Bödeker B, Baumbach JI Volatile organic compounds in exhaled breath of patients with COPD ± lung cancer and their correlation with FEV1-values. Eur Respir J 2014; 44: Suppl 58, P987
- [Background] Westhoff M, Friedrich M, Baumbach JI. Simultaneous measurement of inhaled air and exhaled breath by double multicapillary column ion-mobility spectrometry, a new method for breath analysis: results of a feasibility study. ERJ Open Res. 2022 Feb 14;8(1):00493-2021. doi: 10.1183/23120541.00493-2021. eCollection 2022 Jan. PMID 35174246
- [Result] Bunkowski A, Bodeker B, Bader S, Westhoff M, Litterst P, Baumbach JI. MCC/IMS signals in human breath related to sarcoidosis-results of a feasibility study using an automated peak finding procedure. J Breath Res. 2009 Dec;3(4):046001. doi: 10.1088/1752-7155/3/4/046001. Epub 2009 Sep 23. PMID 21386194
- [Result] Westhoff M, Litterst P, Freitag L, Urfer W, Bader S, Baumbach JI. Ion mobility spectrometry for the detection of volatile organic compounds in exhaled breath of patients with lung cancer: results of a pilot study. Thorax. 2009 Sep;64(9):744-8. doi: 10.1136/thx.2008.099465. Epub 2009 Jan 21. PMID 19158121
- [Result] Westhoff M, Litterst P, Freitag L, Baumbach JI. Ion mobility spectrometry in the diagnosis of sarcoidosis: results of a feasibility study. J Physiol Pharmacol. 2007 Nov;58 Suppl 5(Pt 2):739-51. PMID 18204189
- [Result] Bunkowski A, Maddula S, Davies AN, Westhoff M, Litterst P, Bödeker B, Baumbach JI. One-year time series of investigations of analytes within human breath using ion mobility spectrometryInt. J. Ion Mobil. Spec. (2010) 13:141-148
- [Result] Westhoff, M, Litterst P, Maddula S, Bödeker B, Rahman S, Davies AN, Baumbach JI. Differentiation of chronic obstructive pulmonary disease (COPD) including lung cancer from healthy control group by breath analysis using ion mobility spectrometry. Int. J. Ion Mobil. Spec. (2010) 13:131-139
- [Result] Vautz W. Baumbach JI, Westhoff M, Züchner, K, Carstens ETH, Perl T. Breath sampling control for medical application. Int. J. Ion Mobil. Spec. (2010) 13:41-46
- [Result] Westhoff M, Rickermann M, Litterst P, Baumbch JI. Exogenous factors of influence on exhaled breath analysis by ion-mobility spectrometry (MCC/IMS) Int J Ion Mobil Spectr 2019, https://doi.org/10.1007/s12127-019-00247-x
- [Result] Westhoff, M., Rickermann, M., Franieck, E. Litterst P, Baumbach JI. Time series of indoor analytes and influence of exogeneous factors on interpretation of breath analysis using ion mobility spectrometry (MCC/IMS). Int. J. Ion Mobil. Spec. (2019) 22: 39. https://doi.org/10.1007/s12127-019-00243-1